CLINICAL TRIAL: NCT00260663
Title: The Hearing Aid Effectiveness After Aural Rehabilitation (HEAR) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SLI 04-265
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2008-01

CONDITIONS: Hearing Loss
Keywords: Hearing Impaired Rehabilitation; Hearing Aids; Randomized Controlled Trials; Cost Effectiveness; Quality of life; Patient Compliance
MeSH Terms: conditions — Hearing Loss; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Group hearing aid fittings; Procedure: Group hearing aid follow-up

INTERVENTIONS:
Procedure: Group hearing aid fittings
Procedure: Group hearing aid follow-up

SUMMARY:
This study compares the effectiveness of hearing aid appointments provided in a group format to those provided in an individual format. We are asking if hearing aid training with group appointments is as good as or better than with individual appointments.

DETAILED DESCRIPTION:
Background: The number of hearing aids dispensed by the VA has nearly quadrupled from 75,000 in 1996 to over 283,000 in 2003. However, the number of audiologists serving this population has less than doubled (72% increase) in the same period. This imbalance has resulted in burgeoning waiting times for audiology appointments, negatively impacting the quality of life of thousands of veterans while they wait for hearing aids. Reduction in waiting times through more efficient use of limited resources while maintaining high quality care is of great interest to VA leadership. Objectives: The orientation portion of the hearing aid fitting appointment and the hearing aid follow-up visit 4 The researcherseks later impart standard information relevant to all new hearing aid patients, and may be highly conducive to group format. Our specific aims are to compare group and the current standard of individual aural rehabilitation appointments to determine if: 1) group visits are at least as effective ('non-inferior') as individual visits for each audiology appointment, and 2) the use of group visits leads to lower costs for the VA. Methods: The researchers propose a non-inferiority, randomized clinical trial to compare the effectiveness of group vs. individual audiology appointments. The researchers will compare group vs. individual visits for two types of audiology appointments: hearing aid fitting (orientation only) and hearing aid follow-up. The researchers hypothesize that: 1) group visits are at least as effective as individual visits, as measured by hearing-related quality of life and hearing aid adherence, and 2) group visits lead to cost savings, not just in the immediate treatment period, but throughout a 6-month aural rehabilitation period. Setting and Population. The researchers propose to enroll 660 new hearing aid patients from the audiology clinics at the Seattle and American Lake Divisions of VA Puget Sound Health Care System. Randomized Interventions. Patients will be randomized to group vs. individual orientation (intervention #1) and group vs. individual follow-up (intervention #2) visits. Status: Recruitment is completed. The primary effectiveness outcome will be hearing-related quality of life 6 months after the hearing aid fitting. Secondary effectiveness outcomes will include hearing aid adherence and satisfaction with hearing amplification. Cost and utilization outcomes will include audiology labor for the initial visits and subsequent unplanned visits, the cost of hearing aids, and the number of hearing aid repairs. The researchers selected a time frame of 6 months because pilot data show that 75% of unplanned visits occur in the first 6 months. Analysis. An intention-to-treat analysis will be used to minimize bias due to subject self-selection. The researchers have chosen a sample size adequate to detect non-inferiority of hearing-related quality of life in patients undergoing group rehabilitation in either intervention. Analyses for each intervention will be stratified by degree of hearing loss, binaural vs. monaural hearing aid use, and group vs. individual appointment of the other intervention. Cost-effectiveness analyses will be pursued if greater effectiveness and higher costs are both documented, in which case pilot calculations of the unit cost to obtain an additional successfully treated patient (those with a clinically important improvement of 6 points on the Inner EAR scale) will be made. Benefit to VA. This proposal directly addresses three of the VA's designated research areas: sensory disorders, aging, and health services. In addition, this application is directly responsive to an HSR&D Solicitation on sensory disorders and loss. This project has the potential to help VA leadership identify more efficient treatment that maintains high quality care for one of the most common disabilities in veterans, and to provide insight into the value of group visits as a model of care.

ELIGIBILITY:
Inclusion Criteria:

New hearing aid users at VA Puget Sound; eligible for VA hearing aids

Exclusion Criteria:

Prior hearing aid users; Inability to participate in a group rehabilitation sessions or to complete follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Hearing-related quality of life, hearing aid adherence

SECONDARY OUTCOMES:
Satisfaction, costs, utilization

CONTACTS AND LOCATIONS:
Overall Officials: Margaret P. Collins, PhD MS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

REFERENCES:
- [Result] Collins MP, Liu CF, Taylor L, Souza PE, Yueh B. Hearing aid effectiveness after aural rehabilitation: individual versus group trial results. J Rehabil Res Dev. 2013;50(4):585-98. doi: 10.1682/jrrd.2012.03.0049. PMID 23934877
- [Result] Liu CF, Collins MP, Souza PE, Yueh B. Long-term cost-effectiveness of screening strategies for hearing loss. J Rehabil Res Dev. 2011;48(3):235-43. doi: 10.1682/jrrd.2010.03.0041. PMID 21480098
- [Result] Collins MP, Souza PE, Liu CF, Heagerty PJ, Amtmann D, Yueh B. Hearing aid effectiveness after aural rehabilitation - individual versus group (HEARING) trial: RCT design and baseline characteristics. BMC Health Serv Res. 2009 Dec 15;9:233. doi: 10.1186/1472-6963-9-233. PMID 20003515
- [Result] Collins MP, Souza PE, O'Neill S, Yueh B. Effectiveness of group versus individual hearing aid visits. J Rehabil Res Dev. 2007;44(5):739-49. doi: 10.1682/jrrd.2007.02.0029. PMID 17943685
- [Result] Yueh B, Shekelle P. Quality indicators for the care of hearing loss in vulnerable elders. J Am Geriatr Soc. 2007 Oct;55 Suppl 2:S335-9. doi: 10.1111/j.1532-5415.2007.01340.x. No abstract available. PMID 17910555
- [Result] Yueh B, Collins MP, Souza PE, Heagerty PJ, Liu CF, Boyko EJ, Loovis CF, Fausti SA, Hedrick SC. Screening for Auditory Impairment-Which Hearing Assessment Test (SAI-WHAT): RCT design and baseline characteristics. Contemp Clin Trials. 2007 May;28(3):303-15. doi: 10.1016/j.cct.2006.08.008. Epub 2006 Aug 30. PMID 17030153